CLINICAL TRIAL: NCT06846047
Title: Therapeutic Effects of Electrical Vestibular Stimulation (EVS) on Balance and Gait
Acronym: VST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neursantys Inc (Industry)
Collaborators: Mitacs (Industry); University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB22-1006_MOD4
Record Dates: First submitted 2025-02-03; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Vestibulopathy
Keywords: age-related balance decline

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Electrical vestibular stimulation treatment (Experimental): Participants in this Arm will receive active treatment with swsEVS applied
  Interventions: Device: electrical vestibular stimulation (EVS)
- Sham stimulation treatment (Sham Comparator): Participants in this Arm will receive sham treatment with no swsEVS applied.
  Interventions: Device: Sham Comparator

INTERVENTIONS:
Device: electrical vestibular stimulation (EVS) — EVS involves electrically activating the vestibular nerves by passing small electrical currents through electrodes placed on the mastoid processes (behind the ears) via battery powered, constant current isolated stimulators.
  Arms: Electrical vestibular stimulation treatment
Device: Sham Comparator — No current is applied during EVS treatment
  Arms: Sham stimulation treatment

SUMMARY:
The aim of the study to is determine the safety, feasibility, efficacy, and persistence of non-invasive EVS to improve balance and gait performance in healthy individuals across the lifespan. Specifically, our objective is to measure balance and gait performance before, during and after exposure to single sessions and across repeated sequences of EVS at multiple study partner sites.

DETAILED DESCRIPTION:
Background and Rationale

Standing balance and stable gait are maintained through the integration of sensory feedback from the visual, somatosensory (muscle, skin, tendon, and joint receptors), and vestibular systems. The quality of this feedback, and the ability of the central nervous system (brain and spinal cord) to integrate these signals and generate appropriate motor responses dictates balance and gait performance. Age-related balance decline, clinically known as presbystasis, is one of the most visible and debilitating signs of aging. More than 60 million people in the U.S. over the age of 40 live with age-related balance impairments that increase their risks of fall-related injuries and make it increasingly difficult to continue living actively and independently. 1-in-3 adults above the age of 65 falls each year and falls are the leading cause of death in seniors. But there are less than 20,000 clinical specialists in the U.S. with the tools to diagnose balance impairments, so for most people, little is done to address declining balance until after a fall-related injury occurs. The solution offered to most older adults is a mechanical balance aid such as a walker, whose prolonged use only further destabilizes balance.

Vestibular dysfunction has been identified as the primary cause of balance decline in more than 55% of adults over age 50, or around 34 million people in the U.S. This dysfunction impacts both the peripheral vestibular organs in the inner ear and central vestibular processing in the brain, and it has also been linked to cognitive decline. Current therapeutic options to restore lost balance function are limited to high-risk surgical vestibular implants. The current standard of care is exercise-based therapy that aims to help compensate for vestibular balance decline, but there remains a critical gap: no widely available non-invasive solution exists to restore lost vestibular function or prevent further deterioration.

A growing body of research indicates that low-level, non-invasive electrical stimulation of the vestibular balance system (EVS) can induce neuroplastic changes at both cellular and circuit levels, effectively restoring peripheral and central vestibular functions. Restored vestibular function has also been linked to restored cognitive function. The investigators have developed a novel sub-threshold wideband stochastic EVS (swsEVS) neuroplastic stimulation, which targets peripheral and central vestibular pathways. Multiple studies have demonstrated that the swsEVS frequencies and current levels are safe, comfortable, well-tolerated, and have no adverse side effects. These studies have also demonstrated that a therapeutic treatment protocol with 18 twenty-minute swsEVS sessions delivered over a 5-6-week period resulted in significant improvements in balance performance in otherwise healthy adults aged 50-98 years old. These improvements are attributed to neuroplastic restoration of both peripheral and central vestibular function. The observed improvements persisted for at least 3-6 months and were sufficient to recategorize high fall risk individuals to lower fall risk.

Objectives

With the proposed pre-clinical study, the investigators aim to determine the safety, feasibility, efficacy, and persistence of the above non-invasive swsEVS to improve balance and gait performance in healthy individuals across the lifespan. Specifically, our objective is to measure balance and gait performance before, during and after exposure to single sessions and across repeated sequences of swsEVS at multiple study partner sites. The investigators predict that swsEVS-induced neuroplasticity may promote recovery of vestibular function via documented mechanisms that include: 1) regeneration of vestibular hair cells; 2) an increase in synaptic gain in the vestibular system, 3) an increase in vestibular afferent/efferent nerve fibre conductivity and excitability, and 4) increased central neural integration of sensory signals (vestibular, visual, somatosensory) for motor control. As such, our main hypothesis with this research is that exposure to repeated sequences of swsEVS will enhance balance and gait performance (e.g., walking cadence, stability, etc.).

A secondary objective of this study is to determine if changes in vestibular function are accompanied by measurable changes in cognitive function.

Finally, a tertiary objective of this research is to determine if swsEVS has any potential benefit for participants suffering from occasional headaches. There is some anecdotal evidence that EVS could help with headaches, particularly for so-called "vestibular migraines"; however, to date this has not been formally studied.

Participants

Healthy young and older adult participants (18 - 100 years of age) will be recruited in this study. Participants will be recruited at each study site from their local community by word of mouth, study ad postings, and the UCalgary Participate website. All participants will be given detailed written and oral explanations of experimental goals and procedures, and the protocol will be approved by UCalgary's Clinical Health Research Ethics Board (CHREB). Participants will provide written informed consent prior to participation.

Methodology

Participation in this experiment will involve 18 testing sessions over a 5-6- week period, as well as 3-week, 6-week, 3-month, and 6-month follow up sessions. Each testing and follow-up session will last under 1-hour. The proposed project will employ six primary techniques: (i) electrical vestibular stimulation (swsEVS); (ii) accelerometry; (iii) smartphone app-based gait and balance tests; (iv) clinician-administered Functional Gait Assessments; (v) static and dynamic balance tests using an instrumented balance platform; (vi) cognitive assessments. swsEVS test administrators will also collect information about any adverse events during each visit and since the last visit. Participants will also complete questionnaires upon entering and exiting the study to assess the prevalence and severity of headaches, cognition, dizziness, level of physical activity, as well as to determine if these headaches are causing any notable disability.

(i) Electrical Vestibular Stimulation (EVS) involves electrically activating the peripheral vestibular system by passing small electrical currents through electrodes placed on the mastoid processes (behind the ears) via battery powered, constant current isolated stimulators. This non-invasive, safe and painless bioelectronic stimulation technique commonly utilizes either a stochastic signal (white noise) or monopolar or bipolar square- or sine-wave pulses. EVS typically used different bandwidths of stimulation, from broad-band (0-1 kHz) to narrow-band (0-2 Hz).EVS may also be applied at different stimulation amplitudes, ranging from those that are below the level of evoking any sensation by the participant ("sub-threshold"; typically < 0.5 mA), to those that evoke overt vestibular sensations and balance responses ("supra-threshold"; > 0.5 mA). The swsEVS neuroplastic restoration in the present study delivers subthreshold, wideband, stochastic stimuli via 2 pairs of disposable single-use electrodes attached to each mastoid and the back of the neck. EVS does not ever exceed +/- 3 mA (hardware and software limited), giving it an excellent safety profile across a large and growing body of scientific literature.

(ii) Accelerometry: Participants will be instrumented with wearable accelerometers (Phybrata Sensor; PROTXX Inc.) on their head over top of the right mastoid process, as well as on the top of each foot. The sensor placed on the head has been validated as a measure of gait and balance performance in multiple previous studies. The sensors placed on the top of the foot will be used to reconstruct step-by-step foot placement kinematics during gait testing. Sensors attached to the head will be affixed to the skin with disposable double-sided medical adhesive tape, after cleaning the skin with an alcohol swab. Sensors applied to the foot during gait testing will be affixed with medical tape. The accelerometers automatically collect and relay the kinematic data to a smartphone app-based system.

(iii) Smartphone App-Based Gait and Balance Testing: Gait and balance assessments will be performed using a smartphone app developed by PROTXX Inc. The app guides the user through the experimental procedures through on-screen instructions and auditory beeps. Investigators will use the app to perform assessments of quiet standing (3 x 2 min intervals of standing still and relaxed with their arms at their sides; 1 min eyes open, 1 min eyes closed), as well as the standard Timed Up and Go (TUG) task and an over-ground walking task. For the TUG task, participants will start seated in a chair, then when prompted by the app, will stand up, walk 3 m forward to a pilon on the floor, turn around 180 degrees, then return to the chair and sit down. For the over-ground walking task, participants will simply start standing with their toes over a tape line on the floor, then they will walk forward (< 50') to an end target pilon.

(iv) Functional Gait Assessment (FGA): The investigators will have trained clinicians administer the FGA, which involves timing 10 different tests of mobility, including: 1) level surface walking (20'), 2) 'change-in-gait-speed' task alternating between 'slow' and 'fast' speeds (5' each), 3) walking with horizontal head turns every 3 steps (20'), 4) walking with vertical head turns every 3 steps (20'), 5) walking with pivot turn to reverse direction and stop (5'), 6) walking with a step over a 9" obstacle (i.e., the height of 2 shoe boxes), 7) walking with narrow base of support (i.e., stepping 'heel-to-toe') for 10 steps, 8) walking with eyes closed (20'), 9) walking backwards (20'), and 10) walking up and down a set of 4 steps, using a railing if necessary.

(v) Cognitive Assessments: Cognitive assessments will utilize paper-based questionnaire forms of the Symbol Digit Matching Task (SDMT) and the Montreal Cognitive Assessment (MoCA).

Experiment Overview

During their initial intake session at the study site, all participants will undergo EVS threshold testing to determine normalized levels of EVS that result in balance perturbations. This EVS threshold testing will be carried out by administering very low currents (starting at ~0.1 mA) to participants standing with their eyes closed and increasing the current level across trials until an EVS balance threshold is determined.

During all 18 subsequent testing sessions, participants will perform gait and balance tests administered via a smartphone app (see below) before and after a single continuous session of swsEVS (<20 min). During each swsEVS session, participants will alternate between sitting, standing on the hard floor, and standing on a foam pad, with intervals of having their eyes open and closed. An investigator will always be nearby the participants to protect them from falling and provide postural support if needed.

Cognitive testing and headache questionnaires will be completed during the first and last of the 18 treatment sessions.

During the 3-week, 6-week, 3-month, and 6-month follow up sessions, participants will repeat gait and balance tests to assess the persistence of any performance improvements measured after the 18 testing sessions.

Statistical Design

To determine the therapeutic efficacy of repeated EVS sessions, dependent variables will be submitted to repeated measures ANCOVA with stimulation type ('sub-threshold', 'supra-threshold') and sex ('male', 'female') as between subject factors, and age as a covariate. Further exploratory analysis of relationships between age and different dependent variables will be performed using Pearson correlations. An alpha level of 0.05 will be used as the statistical significance threshold for all testing.

ELIGIBILITY:
Inclusion Criteria:

1. Able to complete balance assessments such as standing with feet together/eyes open and feet together/eyes closed, both for at least 1 minute at a time, with no more than 1 minute rest required between tests.
2. Able to complete gait assessment tests such as walking up to 200m on a flat surface without assistance.

Exclusion Criteria:

1. Participants must not be using a pacemaker, cochlear implant, or any other implanted electronic device.
2. Participants must be free from any diagnosed neurological or musculoskeletal injuries and/or disorders other than those explicitly being investigated (i.e., vertigo, multiple sclerosis, Parkinson's disease, concussion).
3. Participants must have the mental capacity to provide consent and perform tasks required by the experiment.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Postural Sway Measure of Balance Performance | From enrollment through the end of treatment and up to 6 months post treatment
  Postural sway will be calculated from acceleration profiles of the head measured using data from a head-mounted accelerometer in eyes open and eyes closed conditions. The raw acceleration signals are in units of G. The outcome measure is expressed as a sway power value (in Watts). Sway power measured during static standing has been shown to be a precise, quickly administered assessment of balance performance with excellent sensitivity in the identification of older adult fallers. We will complete the above 2-minute postural sway assessment (60 seconds eyes open followed by 60 seconds eyes closed) immediately before and after each of the 18 EVS treatment sessions in order to track each study participant's changes in balance performance following each treatment session and the cumulative change following completion of the 18 session treatment protocol.
Sensory Integration Measure of Balance Performance | From enrollment through the end of treatment and up to 6 months post treatment
  Sensory integration will be calculated from acceleration profiles of the head measured using data from a head-mounted accelerometer in eyes open and eyes closed conditions. The raw acceleration signals are in units of G. The outcome measure is calculated using a frequency spectrum analysis of the normalized contributions of the three sensory inputs (visual, vestibular, proprioceptive) to balance control. Sensory integration measured during static standing using wearable sensors or computerized dynamic posturography has been shown to be a precise, quickly administered assessment of sensory contributions to balance control with excellent sensitivity in the identification of sensory impairments that disrupt balance in older adults. Sensory reweighting will be calculated using the head acceleration data from the above 2-minute postural sway assessment (60 seconds eyes open followed by 60 seconds eyes closed) immediately before and after each of the 18 EVS treatment sessions in order to tr
Gait Velocity Measure of Gait Performance | From enrollment through the end of treatment and up to 6 months post treatment
  Dynamic gait performance will be measured using data from a head-mounted accelerometer. The raw acceleration signals are in units of G. For dynamic gait tasks, the outcome measures will be the peak walking speed (in Meters per Second) achieved over a set of pre-defined distances from 3 meters to 100 meters. Wearable sensor-based gait velocity tests are widely used in research for older adults with and without pathology, and have norm referenced values and robust clinimetric properties. The above gait velocity measurements will be carried out prior to the first EVS treatment session and following the final (18th) EVS treatment session in order to track the cumulative change in each study participant's gait performance following completion of the 18 session treatment protocol.
Gait Cadence Measure of Gait Performance | From enrollment through the end of treatment and up to 6 months post treatment
  Dynamic gait performance will be measured using data from a head-mounted accelerometer. The raw acceleration signals are in units of G. For dynamic gait tasks, the outcome measures will be gait cadence (in Steps per Second) over a set of pre-defined distances from 3 meters to 100 meters. Wearable sensor-based gait cadence tests are widely used in research for older adults with and without pathology, and have norm referenced values and robust clinimetric properties. The above gait cadence measurements will be carried out prior to the first EVS treatment session and following the final (18th) EVS treatment session in order to track the cumulative change in each study participant's gait performance following completion of the 18 session treatment protocol.
Step Length Measure of Gait Performance | From enrollment through the end of treatment and up to 6 months post treatment
  Dynamic gait performance will be measured using data from a head-mounted accelerometer. The raw acceleration signals are in units of G. For dynamic gait tasks, the outcome measures will be step length (in Meters) over a set of pre-defined distance from 3 meters to 100 meters. Wearable sensor-based step length tests are widely used in research for older adults with and without pathology, and have norm referenced values and robust clinimetric properties. The above step length measurements will be carried out prior to the first EVS treatment session and following the final (18th) EVS treatment session in order to track the cumulative change in each study participant's gait performance following completion of the 18 session treatment protocol.
Step Trajectory Measure of Gait Performance | From enrollment through the end of treatment and up to 6 months post treatment
  Dynamic gait performance will be measured using data from a head-mounted accelerometer. The raw acceleration signals are in units of G. For dynamic gait tasks, the outcome measures will be the distribution of head trajectories during each step (in Angular Degrees) over a set of pre-defined distances from 3 meters to 100 meters. Wearable sensor-based step trajectory tests are widely used in research for older adults with and without pathology, and have norm referenced values and robust clinimetric properties. The above step trajectory measurements will be carried out prior to the first EVS treatment session and following the final (18th) EVS treatment session in order to track the cumulative change in each study participant's gait performance following completion of the 18 session treatment protocol.

SECONDARY OUTCOMES:
Symbol Digit Matching Task (SDMT) Measure of Cognitive Performance | From enrollment through the end of treatment and up to 6 months post treatment
  This secondary outcome variable will measure changes in cognitive performance scores before vs. after the 18-session EVS intervention period of the study. For assessment of cognitive performance, the measurement scale will be the Symbol Digit Matching Task (SDMT). SDMT quantifies the number of symbol-digit matching pairs the participant completes in 90 seconds.
Montreal Cognitive Assessment (MoCA) of Cognitive Performance | From enrollment through the end of treatment and up to 6 months post treatment
  This secondary outcome variable will measure changes in cognitive performance scores before vs. after the 18-session EVS intervention period of the study. For assessment of cognitive performance, the measurement scale will be the Montreal Cognitive Assessment (MoCA). The MoCA is scored on a 0 to 30 scale.

OTHER OUTCOMES:
Migraine Disability Assessment (MIDAS) of Headaches | From enrollment through the end of treatment and up to 6 months post treatment
  For participants suffering from headaches, this tertiary outcome variable will determine if there are any changes after vs. before the 18-session EVS intervention period. For assessments of headaches, the measurement scales will be the Migraine Disability Assessment (MIDAS). The MIDAS is scored by totaling the number of days indicated by the user across a 5-item questionnaire.
Dizziness Handicap Inventory (DHI) of Dizziness | From enrollment through the end of treatment and up to 6 months post treatment
  For participants suffering from dizziness, this tertiary outcome variable will determine if there are any changes after vs. before the 18-session EVS intervention period. For assessments of dizziness, the measurement scale will be the Dizziness Handicap Inventory (DHI). The DHI is scored by totaling the value indicated by the subject (0 = No, 2 = Sometimes, 3 = Always) across a 25-item questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan M Peters, PhD, Principal Investigator — University of Calgary
Locations (4):
- United States (2):
  - Caring Hands Caregivers, Cupertino, California
  - Neursantys, Menlo Park, California
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - Sparx Wellness Institute, Dieppe, New Brunswick

IPD SHARING:
Plan to Share IPD: Yes
de-identified balance and gait performance data
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Start date: March 1, 2027 End date: March 1, 2029
Access Criteria: Study participants and other research groups studying age-related balance decline.

REFERENCES:
- [Background] Ralston JD, Raina A, Benson BW, Peters RM, Roper JM, Ralston AB. Physiological Vibration Acceleration (Phybrata) Sensor Assessment of Multi-System Physiological Impairments and Sensory Reweighting Following Concussion. Med Devices (Auckl). 2020 Dec 8;13:411-438. doi: 10.2147/MDER.S279521. eCollection 2020. PMID 33324120
- [Background] 13. King J, Walters N, Clark S, Mehri N, Al Bastami J, Chan A, Ferrier E, Rodrigues N, Rempel J, Ralston JD, Peters RM. "Electrical Vestibular Stimulation for Therapeutic Balance Enhancement in Older Adults". Submitted for publication, 2024.
- [Background] 12. Ralston JD, King JA, Rempel J, Peters RM, Chima B. "PHYBRATA Biomarker Assessments of Age-Related Balance Impairments and EVS Balance Restoration." 2023 Biomarkers of Aging Symposium, Buck Institute for Research on Aging, Novato, California, USA, Dec 4, 2023.
- [Background] 11. King JA, Banman CJ, Walters N, Clark S, Ralston JD, Peters RM. "Electrical Vestibular Stimulation Therapeutics for Balance and Gait in Older Adults." Canadian Association on Gerontology 52nd Annual Scientific and Educational Meeting, CAG2023, Toronto, Ontario, Canada, October 26-28, 2023.
- [Background] 10. Ralston JD, King J, Rempel J, Peters RM. "Wearable Bioelectronic Balance Restoration in Older Adults." AGE-WELL Annual Conf, Toronto, Ontario, Oct 24-26, 2023.
- [Background] Dilda V, MacDougall HG, Curthoys IS, Moore ST. Effects of Galvanic vestibular stimulation on cognitive function. Exp Brain Res. 2012 Jan;216(2):275-85. doi: 10.1007/s00221-011-2929-z. Epub 2011 Nov 11. PMID 22076407
- [Background] Lopez C, Cullen KE. Electrical stimulation of the peripheral and central vestibular system. Curr Opin Neurol. 2024 Feb 1;37(1):40-51. doi: 10.1097/WCO.0000000000001228. Epub 2023 Oct 25. PMID 37889571
- [Background] Pires APBA, Silva TR, Torres MS, Diniz ML, Tavares MC, Goncalves DU. Galvanic vestibular stimulation and its applications: a systematic review. Braz J Otorhinolaryngol. 2022 Nov-Dec;88 Suppl 3(Suppl 3):S202-S211. doi: 10.1016/j.bjorl.2022.05.010. Epub 2022 Jul 5. PMID 35915031
- [Background] Dlugaiczyk J, Gensberger KD, Straka H. Galvanic vestibular stimulation: from basic concepts to clinical applications. J Neurophysiol. 2019 Jun 1;121(6):2237-2255. doi: 10.1152/jn.00035.2019. Epub 2019 Apr 17. PMID 30995162
- [Background] Deveze A, Bernard-Demanze L, Xavier F, Lavieille JP, Elziere M. Vestibular compensation and vestibular rehabilitation. Current concepts and new trends. Neurophysiol Clin. 2014 Jan;44(1):49-57. doi: 10.1016/j.neucli.2013.10.138. Epub 2013 Nov 6. PMID 24502905
- [Background] Smith PF. Aging of the vestibular system and its relationship to dementia. Curr Opin Neurol. 2024 Feb 1;37(1):83-87. doi: 10.1097/WCO.0000000000001231. Epub 2023 Nov 30. PMID 38038627
- [Background] 3. Agrawal Y, Smith PF, Merfeld DM, "6.36 - Dizziness, Imbalance and Age-Related Vestibular Loss, Editor(s): Bernd Fritzsch, The Senses: A Comprehensive Reference (Second Edition)." Elsevier,2020, p. 567-580, ISBN 9780128054093.
- [Background] Iwasaki S, Yamasoba T. Dizziness and Imbalance in the Elderly: Age-related Decline in the Vestibular System. Aging Dis. 2014 Feb 9;6(1):38-47. doi: 10.14336/AD.2014.0128. eCollection 2015 Feb. PMID 25657851
- [Background] Davis LE. Dizziness in elderly men. J Am Geriatr Soc. 1994 Nov;42(11):1184-8. doi: 10.1111/j.1532-5415.1994.tb06986.x. PMID 7963205
- [Derived] King JA, Walters N, Rodrigues N, Al Bastami J, Mehri N, Chan A, Spencer M, Clark S, Ferrier E, Orr SL, Rempel J, Hauenstein A, Roper JM, Ralston JD, Peters RM. Electrical vestibular stimulation to improve balance in older adults: a pilot randomized controlled trial. J Neuroeng Rehabil. 2025 Oct 31;22(1):231. doi: 10.1186/s12984-025-01749-y. PMID 41174737